CLINICAL TRIAL: NCT00355368
Title: Phase 4 Study of Succinylcholine Versus Rocuronium as Neuromuscular Blocking Agent for Emergency Intubation in Intensive Care
Brief Title: Succinylcholine Versus Rocuronium for Emergency Intubation in Intensive Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Stephan Marsch, Professor and Chairman of Medical ICU, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK 145/05
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Results first posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-11

CONDITIONS: Intubation
Keywords: intubation; intensive care; neuromuscular depolarizing agents; neuromuscular nondepolarizing agents; neuromuscular blocking agents
MeSH Terms: interventions — Succinylcholine; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Succinylcholine (Active Comparator)
  Interventions: Drug: Succinylcholine
- Rocuronium (Active Comparator)
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Succinylcholine — 1mg/kg iv
  Arms: Succinylcholine
Drug: Rocuronium — 0.6mg/kg iv
  Arms: Rocuronium

SUMMARY:
Emergency intubation of patients in intensive care is a high-risk endeavour. For many decades, succinylcholine has been the neuromuscular blocking agent of choice. However, succinylcholine may have life-threatening side effects and is contraindicated in a variety of diseases relevant in intensive care. The nondepolarizing agent rocuronium has been propagated as alternative for succinylcholine. Though a recent meta-analysis found no difference in intubating conditions between succinylcholine and rocuronium in elective cases, there are no data in emergent cases in intensive care. The aim of the present study is to compare succinylcholine and rocuronium with regard to 1) quality of intubating conditions, 2) length of the intubating sequence, 3) failed intubating attempts, 4) hemodynamic sequelae of intubation, and 5) desaturations.

DETAILED DESCRIPTION:
Objective: to compare succinylcholine and rocuronium with regard to 1) quality of intubating conditions, 2) length of the intubating sequence, 3) failed intubating attempts, 4) hemodynamic sequelae of intubation, and 5) desaturations.

Design: prospective, randomized, single-blind study. Setting: Intensive care units of an University Hospital. Patients: adult patients in intensive care requiring emergency intubation. Randomization: 1:1 randomization to either succinylcholine (1mg/kg) or rocuronium (0.6 mg/kg).

Data: 1) assessment of the quality of intubating conditions by means of a score, 2) length of the intubating sequence defined as time between injection of neuromuscular blocking agent and first end-tidal CO2 on the monitor, 3) number of failed intubating attempts, 4) hemodynamic sequelae of intubation, defined as events requiring injection of vasoactive drugs, and 5) desaturations, defined as saturation below 90% and/or any decrease in saturation of 5% or more.

ELIGIBILITY:
Inclusion Criteria:

* indication for emergency intubation in intensive care
* availability of qualified study physician

Exclusion Criteria:

* contraindication against succinylcholine or rocuronium
* indication for awake fibreoptic intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Siegemund, MD, Principal Investigator — Department of Surgical Intensive Care, University of Basel; Stephan C Marsch, MD, DPhil, Principal Investigator — Department of Medical Intensive Care, University of Basel
Locations (1):
- Department of Medical Intensive Care; University of Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Sluga M, Ummenhofer W, Studer W, Siegemund M, Marsch SC. Rocuronium versus succinylcholine for rapid sequence induction of anesthesia and endotracheal intubation: a prospective, randomized trial in emergent cases. Anesth Analg. 2005 Nov;101(5):1356-1361. doi: 10.1213/01.ANE.0000180196.58567.FE. PMID 16243994
- [Derived] Marsch SC, Steiner L, Bucher E, Pargger H, Schumann M, Aebi T, Hunziker PR, Siegemund M. Succinylcholine versus rocuronium for rapid sequence intubation in intensive care: a prospective, randomized controlled trial. Crit Care. 2011 Aug 16;15(4):R199. doi: 10.1186/cc10367. PMID 21846380

RESULTS

PARTICIPANT FLOW:
Groups:
- Succinylcholine: 1mg/kg
- Rocuronium: 0.6mg/kg
Period: Overall Study
Arm/Group | Succinylcholine | Rocuronium
Started | 210 | 210
Completed | 200 | 201
Not Completed | 10 | 9
Not completed — Protocol Violation | 8 | 7
Not completed — cardiac arrest prior to intubation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Succinylcholine | Rocuronium | Total
Number analyzed (Participants) | 210 | 210 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 123 | 108 | 231
  >=65 years | 87 | 102 | 189
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (16) | 63 (14) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 93 | 184
  Male | 119 | 117 | 236
Region of Enrollment [Number; unit: participants]
  Switzerland | 210 | 210 | 420

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Exhibiting Desaturation >5%
Description: decrease of >5% in oxygen saturation measured continuously using pulse oxymetry
Time Frame: at any time between the start of the intubation sequence and 2min after the completion of intubation
Population: ITT
Measure: Number; unit: participants
Arm/Group | Succinylcholine | Rocuronium
Number analyzed (Participants) | 200 | 200
participants | 73 | 66

2. Secondary Outcome: Haemodynamic Sequelae of Intubation
Description: any new haemodynamic alteration requiring immediate intervention
Time Frame: between start of induction sequence and 5 min after completion of intubation
Reporting Status: Not Posted
Measure: Number; unit: participants

3. Secondary Outcome: Time to Completion of Intubation
Description: time interval between the injection of the induction agent and the first appearance of endtidal CO2
Time Frame: time interval between the injection of the induction agent and the first appearance of endtidal CO2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Succinylcholine | Rocuronium
Number analyzed (Participants) | 200 | 200
seconds | 81 (38) | 95 (48)

4. Secondary Outcome: Quality of Intubation Conditions Using a Validated Score: Viby-Mogensen et al. Good Clinical Research Practice (GCRP) in Pharmacodynamic Studies of Neuromuscular Blocking Agents. Acta Anaesthesiol Scand 1996;40:59-74.
Description: The factors laryngoscopy, vocal cords, and response to intubation are individually rated with a score from 1 (bad intubation conditions)to 3 (excellent intubation conditions)and the resulting three scores are summed up. The maximum score is thus 9 while the minimum score is 3.
  Units: measure on a scale
Time Frame: during laryngoscopy and the first minute after completion of intubation
Measure: Mean (Standard Deviation); unit: score points
Arm/Group | Succinylcholine | Rocuronium
Number analyzed (Participants) | 200 | 200
score points | 8.3 (0.8) | 8.2 (0.9)

5. Secondary Outcome: Number of Participants With an Failed First Intubation Attempts
Description: defined as either uncompleted intubation attempt within 90 sec or starting a second intubation attempt
Time Frame: within the first 90 sec following the start of induction
Measure: Number; unit: participants
Arm/Group | Succinylcholine | Rocuronium
Number analyzed (Participants) | 200 | 200
participants | 32 | 36

ADVERSE EVENTS:
Arm/Group | Succinylcholine | Rocuronium
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/210
Other Adverse Events (participants affected / at risk) | 0/210 | 0/210

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes